CLINICAL TRIAL: NCT06644456
Title: Relationship Between CAT Score and Airway Limitation in Adult Smokers
Brief Title: CAT Score and Airway Limitation in Adult Smokers
Acronym: CAT
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Sabri Serhan OLCAY, Assistant Professor, Muğla Sıtkı Koçman University
Other Study IDs: CAT24
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Smokers
Keywords: smoker; CAT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Smokers with airway limitation: Smokers with FEV1<80%
- Smokers without airway limitation: smokers with FEV1>80

SUMMARY:
This study aimed to show the relationship between CAT Score and airway limitation in smokers who applied to MSKU Chest Diseases Polyclinic with respiratory complaints (shortness of breath, cough, sputum, etc.) and underwent respiratory function tests. CAT Score is a measurement used to evaluate the quality of life of Chronic Obstructive Pulmonary Disease (COPD) patients. CAT Score is a scale used to assess patients' symptoms (such as shortness of breath, cough, and sputum) and problems affecting their daily activities. CAT Score usually takes a value between 0 and 40, and a high score may indicate that the patient's quality of life is low. There are studies on the usability of CAT Score in Bronchiectasis, Tuberculosis, and Asthma Diseases other than COPD. We hypothesize that there is a positive correlation between CAT Score and airway limitation in smokers before COPD develops. The study was planned as cross-sectional. Between July 2024 and December 2024, patients who apply to MSKU Chest Diseases Polyclinic with respiratory complaints and have a history of smoking will have their CAT scores, 6-minute walking test, and height and weight measurements performed and recorded. In our study, the comparison of CAT Scores of individuals who smoke and have normal respiratory function test parameters with those who are not normal but excluded from COPD is planned as the primary endpoint, and comparisons of CAT Scores with exercise capacities and body mass indexes are planned as the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history Being over 18 years old Being symptomatic

Exclusion Criteria:

* Having a diagnosis of chronic respiratory disease (COPD, Asthma, IPF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to MSKU Chest Diseases Polyclinic with respiratory complaints and had a history of smoking were subjected to respiratory function tests.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
CAT | day 1
  In our study, the primary endpoint was to compare the CAT scores of individuals who smoked and had normal pulmonary function test parameters with those who were not normal but excluded from COPD.

SECONDARY OUTCOMES:
6MWT-BMI | day 1
  Comparisons of exercise capacities and body mass indexes with CAT Scores are planned as secondary endpoints. Weight and height will be combined to report BMI in kg/m^2. 6mwt distance will be reported as meter

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla EAH, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided